CLINICAL TRIAL: NCT06149351
Title: Determination of the Physiological Profile and Evaluation of the Effect of Intense Physical Exertion Among Professional Athletes
Brief Title: Salivary Biomarkers for Concussion
Acronym: SportCo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sys2Diag (Other Government)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Principal Investigator, Thi Nhu Ngoc VAN, Senior Researcher/Project Manager, Sys2Diag
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-A00188-37; 23.00930.000169 (Other: Comité de protection des personnes (French Ethics committee))
Record Dates: First submitted 2023-11-16; First posted 2023-11-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Sport Related Concussion
Keywords: Concussion, Biomarkers, Sport
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sub-group S-P (Other): 30 professional athletes whose weekly sport practice is more than 8 hours of contact sport.
  Interventions: Diagnostic Test: Bio-fluid analysis for the implementation of a diagnostic test for sport related concussion
- Sub-group S-L (Other): 30 amateur athletes, having moderate physical activity whose weekly sport practice is between 4 and 8 hours of contact sport.
  Interventions: Diagnostic Test: Bio-fluid analysis for the implementation of a diagnostic test for sport related concussion
- Sub-group S-O (Other): 20 control subjects who are occasional sport practitioners, having a low intensity physical activity with weekly practicing time is below 4h, excluding contacted sports.
  Interventions: Diagnostic Test: Bio-fluid analysis for the implementation of a diagnostic test for sport related concussion

INTERVENTIONS:
Diagnostic Test: Bio-fluid analysis for the implementation of a diagnostic test for sport related concussion — Saliva of participants will be sampled for analysis of biomarkers of interest (nucleic acids and proteins). The nucleic acids biomarkers will be quantified by reverse transcription followed by amplification (RT-PCR) and Next Generation Sequencing (NGS) techniques while enzymatic assay methods (ELISA) methods will be used to quantify protein biomarkers.

SUMMARY:
Recently, several salivary biomarkers (proteins and nucleic acids) of sport related concussion have been identified in professional athletes. However, their reference values have not been determined with sufficient robustness to enable their employment in concussion diagnostic tests. Toward a proper interpretation of the signal for a reliable diagnostic test, we aim to evaluate the physiological variations as well as the effect of different intensive trainings on the profile of these salivary biomarkers in professional athletes. Data generated form such analysis will help establish a baseline profile for these biomarkers whose change in intensity associated with concussion could be diagnosed in the future.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged between 18 and 50 years old.
* Participants willing to comply with the study procedures.
* Participants capable of understanding the purpose, nature, and methodology of the study.
* Participants affiliated to a French social security system or beneficiaries of such a system.
* Participants who have signed the non-opposition form to participate in the research.

Non-inclusion Criteria:

* Participant not affiliated to a French social security system or not a beneficiary of such a system.
* Participants deprived of liberty, protected adults, vulnerable individuals, or minors.
* Participants with a proven or suspected chronic infectious disease that may introduce a risk of contamination during sample handling (laboratories not equipped to handle this type of sample).
* Refusal to sign the non-opposition form to participate in the research.

Non-inclusion specific criteria

* Subject who has had a recent stroke or epilepsy event (within the past two months).
* Subject suffering from neurological diseases.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2027-12-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the baseline level of salivary molecular biomarkers | 3 years
  Quantification of salivary small non coding RNA (sncRNA) biomarkers of all study subjects: before, during and after intense or moderate sports practice (training and/or matches).
  Expression level of acid nucleic biomarkers are measured in copies/µL, number of read and fold change.
Evaluate the baseline level of salivary molecular biomarkers | 3 years
  Quantification of salivary biomarkers including ubiquitin c-terminal hydrolase L1 (UCH-L1), glial fibrillary acidic protein (GFAP) and neuron-specific enolase (NSE) proteins of all study subjects: before, during and after intense or moderate sports practice (training and/or matches). Expression level of protein biomarkers including UCL-L1, GFAP, NSE are measured in pg/mL.

SECONDARY OUTCOMES:
Differential analysis of expression signatures of salivary sncRNAs of the three groups | 3 years
  Comparison of expression signatures of salivary sncRNAs among the professional athletes, amateur athletes, and occasional sport practitioners.
  Expression level of acid nucleic biomarkers are measured in copies/µL and fold change.
Differential analysis of expression level of salivary UCH-L1, GFAP, NSE proteins of the three groups | 3 years
  Comparison of expression signatures of salivary UCH-L1, GFAP, NSE proteins among the professional athletes, amateur athletes, and occasional sport practitioners.
  Expression level of protein biomarkers including UCL-L1, GFAP, NSE are measured in pg/mL.
Differential analysis of expression signatures of salivary sncRNAs of the three groups throughout different sport situations | 3 years
  Comparison of expression signatures of salivary sncRNAs before, during and after different training sessions (bodybuilding, contact, etc) and matches.
  Expression level of acid nucleic biomarkers are measured in copies/µL, number of read and fold change.
Differential analysis of expression level of salivary UCH-L1, GFAP, NSE proteins of the three groups throughout different sport situations | 3 years
  Comparison of expression level of salivary UCH-L1, GFAP, NSE proteins before, during and after different training sessions (bodybuilding, contact, etc) and matches.
Differential analysis of expression signatures of salivary sncRNAs of the three groups throughout the sports season | 3 years
  Comparison of expression signatures of salivary sncRNAs at the beginning, in the middle and by the end of the sports season.
  Expression level of acid nucleic biomarkers are measured in copies/µL, number of read and fold change.
Differential analysis of expression level of salivary UCH-L1, GFAP, NSE proteins of the three groups throughout the sports season | 3 years
  Comparison of expression level of salivary UCH-L1, GFAP, NSE proteins at the beginning, in the middle and by the end of the sports season.
  Expression level of protein biomarkers including UCL-L1, GFAP, NSE are measured in pg/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Thi Nhu Ngoc VAN, Phd, Principal Investigator — Sys2Diag
Locations (1):
- Sys2Diag - Umr9005 Cnrs/Alcen, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Pietro V, Ragusa M, Davies D, Su Z, Hazeldine J, Lazzarino G, Hill LJ, Crombie N, Foster M, Purrello M, Logan A, Belli A. MicroRNAs as Novel Biomarkers for the Diagnosis and Prognosis of Mild and Severe Traumatic Brain Injury. J Neurotrauma. 2017 Jun 1;34(11):1948-1956. doi: 10.1089/neu.2016.4857. Epub 2017 Apr 10. PMID 28279125
- [Background] Di Pietro V, O'Halloran P, Watson CN, Begum G, Acharjee A, Yakoub KM, Bentley C, Davies DJ, Iliceto P, Candilera G, Menon DK, Cross MJ, Stokes KA, Kemp SP, Belli A. Unique diagnostic signatures of concussion in the saliva of male athletes: the Study of Concussion in Rugby Union through MicroRNAs (SCRUM). Br J Sports Med. 2021 Dec;55(24):1395-1404. doi: 10.1136/bjsports-2020-103274. Epub 2021 Mar 23. PMID 33757972